CLINICAL TRIAL: NCT02530177
Title: A Prospective, Longitudinal Study of Chemotherapy-Induced Hair Changes and Alopecia, Skin Aging and Nail Changes in Women With Non-Metastatic Breast Cancer
Brief Title: Study of Chemotherapy-Induced Hair Changes and Alopecia, Skin Aging and Nail Changes in Women With Non-Metastatic Breast Cancer
Status: Active, not recruiting | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: University of Chicago (Other); New York University (Other)
Responsible Party: Sponsor
Other Study IDs: 15-198
Record Dates: First submitted 2015-08-19; First posted 2015-08-20 (Estimated); Last update posted 2025-12-04 (Actual); Status verified 2025-12

CONDITIONS: Non-Metastatic Breast Cancer
Keywords: Alopecia; Skin Aging; Nail Changes; Hair Changes; 15-198
MeSH Terms: conditions — Alopecia | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — saliva (baseline only)

GROUPS / COHORTS (3):
- Patients having CYTOTOXIC CHEMOTHERAPY: Participants will undergo study related assessments and the appropriate HRQoL questionnaires will be administered. Baseline and follow-up clinical assessments will be performed, preferably when the patient presents to the clinic for (clinically indicated) standard-of-care visits. Initially, these visits will be coinciding with the appropriate chemotherapy dosing cycles (as applicable to select study cohorts), and subsequently they will be performed during the standard-of-care follow-up visits.
  Interventions: Other: Clinical Assessments; Behavioral: Questionnaires; Other: Saliva sample
- Patients having ENDOCRINE THERAPY: Participants will undergo study related assessments and Medical and Personal History Questionnaire data collection forms and the appropriate HRQoL questionnaires, will be administered. Baseline and follow-up clinical assessments will be performed, preferably when the patient presents to the clinic for standard-of-care visits. Initially, these visits will be coinciding with the appropriate therapy and subsequently they will be performed during the standard-of-care follow-up visits.
  Interventions: Other: Clinical Assessments; Behavioral: Questionnaires; Other: Saliva sample
- COMPARATOR (menopausal women): Menopausal women will include unrelated visitors accompanying breast cancer patients (e.g. friends) attending the breast medicine or dermatology clinics, or female employees of MSKCC. There will be no follow-up visits (after baseline) for participants in the comparator cohort.
  Interventions: Other: Clinical Assessments; Behavioral: Questionnaires; Other: Saliva sample

INTERVENTIONS:
Other: Clinical Assessments
Behavioral: Questionnaires
Other: Saliva sample — (only once, preferably at baseline)

SUMMARY:
The purpose of this study is to see how many patients develop hair, skin and nail changes due to cancer treatments. The investigators would like to study the clinical factors, genetic markers, and impact on patients' health-related quality of life to learn more about who is at greater risk. We trust that the study will improve our understanding of how cancer patients feel about their skin, hair, and nail conditions. This information will help us determine the burden on breast cancer patients and survivors. It will also help us learn how to prevent these conditions and it may improve the way we treat them and counsel patients.

ELIGIBILITY:
Inclusion Criteria:

* Women newly diagnosed with non-metastatic breast cancer (stage 0-III, any receptor type) at the time of starting chemotherapy (dd-AC-T, CMF, Newer Combination Regimens) or endocrine therapy (tamoxifen, anastrozole, letrozole, exemestane)
* Women ≥ 18 years at the time of enrollment into the study
* Able to communicate in English and participate in the informed consent process
* Able to comply with the follow-up visits, assessments, answering questionnaires

Exclusion Criteria:

* Metastatic breast cancer
* Follow-up care/visits not scheduled at MSKCC
* Any current alopecia especially due to an active scalp and/or hair disorder (e.g. alopecia areata), or a pre-existing condition with sequelae (e.g. scarring alopecia)
* Currently active or uncontrolled medical condition [e.g. thyroid disorder, auto-immune connective tissue disease (e.g. SLE), BMT complications (GVHD)] or medication intake (e.g. HRT), affecting scalp hair
* Prior systemic treatment for any malignancy
* Active secondary cancer requiring cytotoxic chemotherapy
* Planned (or a history of) radiation therapy to the head
* Vulnerable populations [e.g. decisionally impaired (cognitive, psychiatric), terminally ill, prisoners], or patients who, in the opinion of the investigator have a condition that precludes their ability to provide an informed consent
* Men

Volunteer Inclusion Criteria:

* Post menopausal women, with menopausal status defined as (per self report):
* Bilateral salpingo-oophorectomy independent of age
* If natural menopause, age ≥ 50 with cessation of menses for at least 12 months
* Or premenopausal women with premenopausal status defined as <53 years of age with no cessation of menses
* Able to communicate in English and participate in the informed consent process
* Able to comply with the baseline assessments and answering questionnaires
* Women >/= 18 years at the time of enrollment into the study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: MSKCC clinics
Sampling Method: Non-Probability Sample
Enrollment: 546 (Estimated)
Dates: Start 2015-08-19 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Incidence of persistent alopecia | 1 year
  as assessed clinically and by phototrichogram assessments, among women exposed to cytotoxic chemotherapy
Incidence of alopecia | 1 year
  as assessed clinically and by phototrichogram assessments, among women exposed to endocrine therapies

CONTACTS AND LOCATIONS:
Overall Officials: Alina Markova, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — https://www.mskcc.org/